CLINICAL TRIAL: NCT02336048
Title: A Multicenter, Double-Blind, Randomized, and Placebo-controlled Phase Ib Study Evaluating the Safety of Adding Tocilizumab to Standard Premedications Prior to Administration of Obinutuzumab in Combination With Chlorambucil in Patients With Previously Untreated B-Cell Chronic Lymphocytic Leukemia and Comorbidities
Brief Title: A Study Evaluating the Safety of Tocilizumab in Addition to Standard of Care Premedication Given Before Obinutuzumab + Chlorambucil in Participants With Untreated B-Cell Chronic Lymphocytic Leukemia (B-CLL) and Comorbidities
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: This study was terminated early because premedication with tocilizumab was unlikely to reduce the risk of IRR.
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BO29448; 2014-004594-16 (EudraCT Number)
Record Dates: First submitted 2015-01-06; First posted 2015-01-12 (Estimated); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: B-Cell Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Chlorambucil; obinutuzumab; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo + Obinutuzumab + Chlorambucil (Active Comparator): Participants will receive placebo and standard premedications on Days 1 and 2 of Cycle 1 (cycle length= 28 days) along with obinutuzumab and chlorambucil administered for 6 cycles.
  Interventions: Drug: Chlorambucil; Drug: Obinutuzumab; Drug: Placebo; Other: Standard Premedication
- Tocilizumab + Obinutuzumab + Chlorambucil (Experimental): Participants will receive tocilizumab and standard premedications on Days 1 and 2 of Cycle 1 (cycle length= 28 days) along with obinutuzumab and chlorambucil administered for 6 cycles.
  Interventions: Drug: Chlorambucil; Drug: Obinutuzumab; Other: Standard Premedication; Drug: Tocilizumab

INTERVENTIONS:
Drug: Chlorambucil — Chlorambucil at a dose of 0.5 milligrams per kilogram (mg/kg) will be administered orally per local prescribing information, on Days 1 and 15 of Cycles 1 to 6.
Drug: Obinutuzumab — Obinutuzumab at a dose of 100 milligrams (mg) as an intravenous (IV) infusion will be administered on Cycle 1 Day 1; 900 mg as IV infusion on Cycle 1 Day 2; 1000 mg as IV infusion on Cycle 1 Days 8 and 15; and 1000 mg as IV infusion on Day 1 of each subsequent cycle for up to 6 cycles.
  Other Names: RO5072759, GA101, Gazya, Gazyvaro
Drug: Placebo — Placebo matching to tocilizumab will be administered as IV infusion on Cycle 1 Day 1 (prior to the first dose of obinutuzumab).
  Arms: Placebo + Obinutuzumab + Chlorambucil
Other: Standard Premedication — Standard-of-care premedication consisting of antipyretic, antihistamine, and corticosteroid will be administered as per United States Package Insert/ Summary of Product Characteristics on Cycle 1 Days 1 and 2 (prior to the first and second dose of obinutuzumab, respectively).
Drug: Tocilizumab — Tocilizumab at a dose of 8 mg/kg or adjusted dose (up to a maximum threshold of 20 mg/kg) will be administered as IV infusion on Cycle 1 Day 1 (prior to the first dose of obinutuzumab).
  Other Names: RO4877533, RoActemra, Actemra
  Arms: Tocilizumab + Obinutuzumab + Chlorambucil

SUMMARY:
This multicenter, double-blind, randomized, placebo-controlled study will evaluate the safety of a single infusion of tocilizumab versus placebo, administered in addition to standard premedications (antipyretic, antihistamine, and corticosteroid) prior to the first infusion of obinutuzumab administered in combination with oral chlorambucil to participants with previously untreated B-CLL who have comorbidities. All eligible participants will be treated with a total of 6 cycles of obinutuzumab + chlorambucil (cycle length = 28 days).

ELIGIBILITY:
Inclusion Criteria:

* Documented cluster of differentiation (CD) 20+ B-CLL according to NCI/IWCLL guideline
* Total Cumulative Illness Rating Scale (CIRS) score greater than (>) 6 and/or creatinine clearance less than (<) 70 milliliters per minute (mL/min)
* Previously untreated chronic lymphocytic leukemia (CLL) requiring treatment according to NCI/IWCLL guidelines who warrant treatment if they have any of the protocol-specified comorbidities
* Life expectancy > 6 months
* Adequate hematological function, unless abnormalities are caused by underlying CLL
* Agreement to use highly effective contraceptive measures per protocol

Exclusion Criteria:

* Any previous CLL treatment
* Documented transformation of CLL to aggressive non-Hodgkin's lymphoma (Richter's transformation)
* Abnormal laboratory test values, unless abnormalities are caused by underlying CLL
* History of progressive multifocal leukoencephalopathy
* Previous treatment with tocilizumab for any indication
* History of severe allergic or anaphylactic reactions to monoclonal antibody therapy
* Known hypersensitivity to any of the study drugs
* History of prior malignancy unless the malignancy has been treated with a curative intent or is in remission without treatment for at least (>/=) 5 years prior to enrollment and with the exception of curatively-treated basal squamous cell carcinoma of the skin, low grade in situ carcinoma of the cervix, or low grade early stage localized prostate cancer treated surgically with curative intent and or ductal carcinoma in situ of the breast treated with lumpectomy alone
* Treatment with glucocorticoids at any dose (except topical formulations) during the 2 weeks prior to the start of Cycle 1 Day 1. Regular treatment with glucocorticoids (> 5 days duration) is also prohibited during the 4-week screening period
* Ongoing treatment with immunosuppressive medications or anti-tumor necrosis factor biologic therapies
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with this protocol or interpretation of results, including significant cardiovascular or pulmonary disease
* Known active or history of recurrent bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) requiring treatment with intravenous (IV) antibiotics or hospitalization within 4 weeks prior to the start of Cycle 1 Day 1
* Active tuberculosis (TB) requiring treatment within 3 years prior to baseline or latent TB diagnosed during screening that has not been appropriately treated
* Vaccination with live or attenuated vaccines within 28 days prior to start of treatment
* Major surgery (within 4 weeks prior to Cycle 1 Day 1), other than for diagnosis
* Positive test results for chronic hepatitis B infection or positivity for hepatitis B core antibody
* Positive test results for hepatitis C
* Known history of human immuno-deficiency virus (HIV) seropositive status
* Positive test results for human T-lymphotropic virus 1 (HTLV 1)
* Pregnant or lactating women
* Participation in another clinical study with drug intervention unless the last dose administered was greater than 5 half-lives of the study product prior to study start
* Any participant actively taking anti-platelet medication or any participant who is fully anticoagulated with warfarin, low-molecular weight heparin or a novel oral anticoagulant including dabigatran, rivaroxiban, epixiban, and similar
* Previous treatment with B-cell depleting agents
* Any inherited bleeding disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-06-26 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2018-09-21 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to approximately 196 days

SECONDARY OUTCOMES:
Percentage of Participants With Infusion-Related Reactions (IRRs) as Assessed by Investigator and Reviewed by Endpoint Adjudication Committee (EAC) | Day 1 (within 24 hours of first obinutuzumab infusion)
Percentage of Participants With IRRs by Severity According to National Cancer Institute Common Terminology Criteria for Adverse Events Version 4.0 (NCI CTCAE v4.0) | Day 1 (within 24 hours of first obinutuzumab infusion)
Percentage of Participants With IRRS >= Grade 3 as assessed by the Investigator and Reviewed by the EAC | Day 1 (within 24 hours of first obinutuzumab infusion)
Number of Interruptions or Administration rate modifications of the First Infusion of Obinutuzumab | Day 1 (within 24 hours of first obinutuzumab infusion)
Percentage of Treatment Discontinuations due to IRR | Day 1 (within 24 hours of first obinutuzumab infusion)
Percentage of Participants With Overall Response as Assessed by Investigator According to NCI/ International Workshop on Chronic Lymphocytic Leukemia (IWCLL) Guidelines | 84 days after last treatment (up to approximately 280 days)
Percentage of Participants With Negative Results for Minimal Residual Disease (MRD) Measured According to NCI/IWCLL Guidelines | 84 days after last treatment (up to approximately 280 days)
Area Under the Serum Concentration-Time Curve From Time Zero to Extrapolated Infinite Time (AUC[0-inf]) of Obinutuzumab | Cycle 1 Day 1 (C1D1), C1D2: Pre-dose (0 hours [hrs]), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1, C6D1: pre-dose (0 hrs); additionally at 3 months after last treatment (9 months) (1 cycle=28 days)
Maximum Observed Serum Concentration (Cmax) of Obinutuzumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1, C6D1: pre-dose (0 hrs); additionally at 3 months after last treatment (9 months) (1 cycle=28 days)
Terminal Half-Life (t1/2) of Obinutuzumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1, C6D1: pre-dose (0 hrs); additionally at 3 months after last treatment (9 months) (1 cycle=28 days)
Area Under the Serum Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC[0-last]) of Obinutuzumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1, C6D1: pre-dose (0 hrs); additionally at 3 months after last treatment (9 months) (1 cycle=28 days)
Total Clearance (CL) of Obinutuzumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1, C6D1: pre-dose (0 hrs); additionally at 3 months after last treatment (9 months) (1 cycle=28 days)
Volume of Distribution (Vd) of Obinutuzumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1, C6D1: pre-dose (0 hrs); additionally at 3 months after last treatment (9 months) (1 cycle=28 days)
AUC(0-inf) of Tocilizumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D1: immediately after tocilizumab infusion (1 hr); C1D3; C1D8, C1D15, C2D1: pre-dose (0 hrs) (1 cycle=28 days)
Cmax of Tocilizumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D1: immediately after tocilizumab infusion (1 hr); C1D3; C1D8, C1D15, C2D1: pre-dose (0 hrs) (1 cycle=28 days)
t1/2 of Tocilizumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D1: immediately after tocilizumab infusion (1 hr); C1D3; C1D8, C1D15, C2D1: pre-dose (0 hrs) (1 cycle=28 days)
AUC(0-last) of Tocilizumab | C1D1, C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D1: immediately after tocilizumab infusion (1 hr); C1D3; C1D8, C1D15, C2D1: pre-dose (0 hrs) (1 cycle=28 days)
Change From Baseline in Interleukin (IL)-6 Level | C1D1: pre-dose (0 hrs) (Baseline), immediately after tocilizumab and obinutuzumab infusion (1 hr, approximately 7 hrs); C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1: pre-dose (0 hrs); C1D3
  1 cycle=28 days
Change From Baseline in Level of Downstream Biomarker of IL-6 Activation: Soluble IL-6 Receptor (sIL-6R) | C1D1: pre-dose (0 hrs) (Baseline), immediately after tocilizumab and obinutuzumab infusion (1 hr, approximately 7 hrs); C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1: pre-dose (0 hrs); C1D3
  1 cycle=28 days
Change From Baseline in Level of Downstream Biomarker of IL-6 Activation: Ferritin | C1D1: pre-dose (0 hrs) (Baseline), immediately after tocilizumab and obinutuzumab infusion (1 hr, approximately 7 hrs); C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1: pre-dose (0 hrs); C1D3
  1 cycle=28 days
Change From Baseline in Level of Downstream Biomarker of IL-6 Activation: C-Reactive Protein (CRP) | C1D1: pre-dose (0 hrs) (Baseline), immediately after tocilizumab and obinutuzumab infusion (1 hr, approximately 7 hrs); C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1: pre-dose (0 hrs); C1D3
  1 cycle=28 days
Change From Baseline in Level of Downstream Biomarker of IL-6 Activation: Soluble Glycoprotein (gp) 130 | C1D1: pre-dose (0 hrs) (Baseline), immediately after tocilizumab and obinutuzumab infusion (1 hr, approximately 7 hrs); C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1: pre-dose (0 hrs); C1D3
  1 cycle=28 days
Change From Baseline in Level of Downstream Biomarker of IL-6 Activation: Serum Amyloid A (SAA) | C1D1: pre-dose (0 hrs) (Baseline), immediately after tocilizumab and obinutuzumab infusion (1 hr, approximately 7 hrs); C1D2: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D8, C1D15, C2D1: pre-dose (0 hrs); C1D3
  1 cycle=28 days
Percentage of Participants With Depletion in Absolute Lymphocyte Count (ALC) | C1D1,C1D2,C1D8,C1D15: pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C1D3; C2D1: Pre-dose (0 hrs), immediately after obinutuzumab infusion (approximately 7 hrs); C3D1,C4D1,C5D1,C6D1: pre-dose (0 hrs) (1 cycle=28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (14):
- Israel (4):
  - Carmel medical center, Haifa
  - Meir Medical Center; Heamatology Dept, Kfar Saba
  - Kaplan Medical Center; Hematology Institute; Hematolgy Institute, Rehovot
  - Ziv Medical Center, Zfat
- Italy (4):
  - A.O. Universitaria S. Martino Di Genova; Ematologia 1, Genoa, Liguria
  - Asst Grande Ospedale Metropolitano Niguarda; Dipartimento Di Ematologia Ed Oncologia, Milan, Lombardy
  - Ospedale Businco; Ematologia, Cagliari, Sardinia
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia; Oncologia Medica, Sant'Andrea Delle Fratte (PG), Umbria
- RECUH, Oncology Centre of Latvia; Clinic of Chemotherapy and Heamatology, Riga, Latvia
- Spain (4):
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Univ. 12 de Octubre; Servicio de Hematologia, Madrid
  - Hospital Universitario Virgen del Rocio; Servicio de Hematologia, Seville
- Barts & London School of Med; Medical Oncology, London, United Kingdom